CLINICAL TRIAL: NCT07300332
Title: The Impact of Hybrid-type High-intensity Interval Training on Vitamin D Metabolism in Adults With Overweight/Obesity
Brief Title: Exercise Training and Vitamin D Metabolism
Acronym: Hybri-D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Dimitrios Draganidis, Assistant Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UTH_2612_8.10.2025
Record Dates: First submitted 2025-12-09; First posted 2025-12-23 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Obesity & Overweight; Vitamin D
Keywords: overweight; obesity; vitamin D; 25-hydroxyvitamin D; high-intensity interval training
MeSH Terms: conditions — Obesity; Overweight | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group will participate in three hybrid-type high-intensity interval training sessions per week over a 12-week period, while receiving a balanced diet
  Interventions: Other: Exercise training
- Control group (Active Comparator): Control group will receive a balanced diet but will not participate in exercise training
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise training — Receive a balanced diet and participate in three hybrid-type high-intensity interval training sessions per week over a 12-week period
  Arms: Exercise group
Other: Control — Receive a balanced diet but abstain from any type of exercise training
  Arms: Control group

SUMMARY:
The prevalence of Vitamin D deficiency is significantly higher in adults with overweight/obesity compared to those with normal body mass index (BMI). The "entrapment" of Vitamin D in adipose tissue due to impaired lipolytic stimulation and/or adipose tissue dysfunction has been proposed as the driving mechanism. Exercise training has been proposed as a promising strategy to increase mobilization of Vitamin D from adipose tissue, given its well described role in stimulating lipolysis. Indeed, a recent study revealed that participation in moderate-intensity cardiovascular type exercise over winter can mitigate the decline in 25-hydroxyvitamin D [25(OH)D] in adults with overweight/obesity, independent of weight loss. The aim of this study is to investigate the impact of hybrid-type high-intensity interval training over winter on vitamin D metabolism, in adults with overweight/obesity.

DETAILED DESCRIPTION:
Thirty adults with overweight/obesity (both males and females) who will meet the inclusion criteria will be randomly assigned to either an Exercise group (n=15) or a Control group (n=15). The Exercise group will participate in three hybrid-type high-intensity interval training sessions per week over a 12-week period, while receiving a balanced diet. The Control group will receive a balanced diet but will not participate in exercise training. Both groups will provide a resting blood sample and undergo assessment of their body composition (via bioelectrical impedance analysis), daily dietary intake (via dietary recalls) and physical activity level (via accelerometry) at baseline (prior to intervention), 6 weeks and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI = 25-35 kg/m2
* Absence of musculoskeletal injuries
* Absence of chronic health-related complications
* Non-smokers

Exclusion Criteria:

* Consumption of Vitamin D supplements
* Consumption of anti-inflammatory drugs, statins and/or steroids

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Change in 25-hydroxyvitamin D concentration | At baseline, 6 weeks and 12 weeks
  25-OH-VD will be quantitatively determined in serum
Change in plasma Vitamin D binding protein concentration | At baseline, 6 weeks and 12 weeks
  Vitamin D binding protein concentration will be determined in plasma
Change in calcium concentration | At baseline, 6 weeks and 12 weeks
  Calcium concentration will be determined in serum
Change in albumin concentration | At baseline, 6 weeks and 12 weeks
  Albumin concentration will be determined in serum
Change in aspartate aminotransferase (SGOT) concentration | At baseline, 6 weeks and 12 weeks
  SGOT concentration will be determined in serum on a Clinical Chemistry analyzer
Change in alanine aminotransferase (SGPT) concentration | At baseline, 6 weeks and 12 weeks
  SGPT concentration will be determined in serum on a Clinical Chemistry analyzer
Change in gamma-glutamyl transferase (γ-GT) concentration | At baseline, 6 weeks and 12 weeks
  γ-GT concentration will be determined in serum on a Clinical Chemistry analyzer

SECONDARY OUTCOMES:
Change in reduced glutathione concentration | At baseline, 6 weeks and 12 weeks
  Reduced glutathione concentration will be determined in blood erythrocytes
Change in oxidized glutathione concentration | At baseline, 6 weeks and 12 weeks
  Oxidized glutathione concentration will be determined in blood erythrocytes
Change in dietary intake | At baseline, 6 weeks and 12 weeks
  Dietary intake habits will be assessed through dietary recalls
Change in physical activity level | At baseline, 6 weeks and 12 weeks
  Physical activity will be assessed via accelerometry
Change in body composition | At baseline, 6 weeks and 12 weeks
  Body composistion will be assessed via bioelectrical impedance analysis (BIA)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Draganidis, PhD, Principal Investigator — University of Thessaly
Locations (1):
- Department of Physical Education and Sport Science, University of Thessaly, Trikala, Karyes, Greece